CLINICAL TRIAL: NCT03844815
Title: Phase 1 Study of Venetoclax in Combination With Decitabine 10-Day Regimen in Subjects With Acute Myeloid Leukemia
Brief Title: Study of Venetoclax in Combination With Decitabine in Subjects With Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB18-1498
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Cycle 1 of Treatment will be Decitabine days 1-10 plus Venetoclax ramp up on days 1-3 followed by Venetoclax target dose on days 4-21
  Cycle 2 of Treatment will be Decitabine days 1-10 plus Venetcolax target dose days 1-21
  During maintenance Decitabine on days 1-5 plus Venetoclax days 1-21
  Interventions: Drug: Decitabine; Drug: Venetoclax

INTERVENTIONS:
Drug: Decitabine — Decitabine will be administered intravenously at a dose of 20mg per day for 10 days during Cycle 1 (28 day cycle)
  Decitabine will be administered intravenously at a dose of 20mg per day for 10 days of Cycle 2 (28 day cycle).
  Decitabine will be administered intravenously at a dose of 20mg per day for 5 days of each 28 day maintenance cycle
Drug: Venetoclax — Venetoclax administered orally on days 1-21 of cycle 1, cycle 2 and maintenance (28 day cycles). Dose levels will be assigned at time of enrollment anywhere from 100mg-400mg. Dose escalation will follow the 3+3 study design.

SUMMARY:
The main purpose of this study is to learn about the safety and tolerability of an experimental drug, Venetoclax, when it is given along with Decitabine in subjects diagnosed with acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Phase 1: Dose Escalation Phase

  1. High risk AML, including any of the following:

     1. Relapsed or refractory disease
     2. TP53 mutant AML
     3. Adverse risk cytogenetics including any of the following: 3 or more abnormalities; deletions involving chromosomes 5, 7, or 17; abnormalities in chromosome 11 involving MLL; t(6;9); inv(3) or t(3;3)
  2. ECOG performance status 0-2
  3. Age 18 years or older
  4. Adequate organ function as defined by all of the following:

     1. Creatinine clearance ≥30 mL/min, determined by the Cockroft-Gault formula, or measured by a 24 hour urine collection
     2. AST and ALT ≤3 x ULN and bilirubin ≤1.5 x ULN (unless considered due to Gilbert's syndrome or of non-hepatic origin i.e. leukemic involvement).
  5. Patients must be at least 2 weeks from major surgery, radiation therapy, or participation in other investigational trials, and must have recovered from clinically significant toxicities related to these prior treatments.
  6. Patients must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the i initiation of any screening or study specific procedures.
  7. Female patients of childbearing potential must have negative results for a pregnancy test
  8. Patients must be willing to use appropriate contraception
* Phase 2: Dose Expansion Phase During the Phase 2 portion of the study, the subject population will be limited to patients with previously untreated AML with a mutation in TP53. All other inclusion criteria described above will apply.

Exclusion Criteria:

- Key exclusion criteria (apply to both Phase 1 and Phase 2 portions of the study):

1. Concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in this protocol
2. Patients suitable for and willing to receive intensive induction chemotherapy
3. Use of investigational agents and/or anticancer therapy within 2 weeks of study entry (with the exception of hydroxyurea, which is permitted before and during Cycle 1 of therapy until D10, at the discretion of the investigator)
4. Prior treatment with venetoclax, decitabine, or azacitidine
5. Diagnosis of acute promyelocytic leukemia
6. Pregnant or breastfeeding patients
7. Patient known to be positive for HIV
8. Known CNS involvement with AML
9. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

   1. Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
   2. Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative-, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate.
   3. An active second cancer that requires treatment within 6 months of study entry
10. Cardiac history including the following:

    1. History of CHF requiring treatment or Ejection Fraction ≤ 50%
    2. Subject has a cardiovascular disability status of New York Heart Association

    Class > 2, defined as:

    i. Cardiac disease in which patients are comfortable at rest but ordinary physical activity ii. Results in fatigue, palpitations, dyspnea, or anginal pain c. Chronic stable angina
11. Treatment with any of the following within 7 days prior to the first dose of study drug:

    1. Steroid therapy for anti-neoplastic intent
    2. Moderate or strong cytochrome P450 3A (CYP3A) inducers
12. Administration or consumption of any of the following within 3 days prior to the first dose of study drug:

    1. Grapefruit or grapefruit products
    2. Seville oranges (including marmalade containing Seville oranges)
    3. Star fruit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
The rate of dose limiting toxicity (DLT) | 24 months
  Determine the rate of subjects who experience a dose limiting toxicity and the maximum tolerable dose

SECONDARY OUTCOMES:
Levels of toxicity with combination regimen | 24 months
  Levels of toxicity experienced with the combination regimen will be reported using data summaries of adverse events, dose limiting toxicity and other safety parameters.
Assessment of Overall Survival | 24 months
  Survival will be measured in months from the date of subject enrollment to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Olatoyosi Odenike, MD, Principal Investigator — University of Chicago
Locations (1):
- University Of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States